CLINICAL TRIAL: NCT04000321
Title: Management of Retained Placenta With Circular Cord Traction for Placenta Delivery- the "Windmill" Technique of Umbilical Cord Traction
Brief Title: Management of Retained Placenta With the "Windmill" Technique of Umbilical Cord Traction
Acronym: Windmill
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Larry Hinkson, Lead Consultant Obstetrics, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA1/037/19
Record Dates: First submitted 2019-06-13; First posted 2019-06-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Placenta; Retention

STUDY DESIGN:
Intervention Model Description: The primary objective of the study is to compare the success rate of removing the placenta in retained placenta pregnencies between the Windmill technique and the control group. Based on this objective, we expected the difference of success rate between groups of 30% (from the previous study, the success rate of the Windmill technique was 86%. The sample size of 35 participants per group will be required to provide 90% power at a 0.05 two-sided significance level.
Masking Description: The primary objective of the study is to compare the success rate of removing the placenta in retained placenta pregnencies between the Windmill technique and the control group. Based on this objective, we expected the difference of success rate between groups of 30% (from the previous study, the success rate of the Windmill technique was 86% . The sample size of 35 participants per group will be required to provide 90% power at a 0.05 two-sided significance level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Windmill group 30 Mins (Experimental): In the Windmill Group, the Windmill technique is carried out after 30 minutes. The windmill technique of the umbilical cord for placental development is performed by a trained obstetrician or midwife with a doctor presence. In a frustrated attempt to develop placenta using the Windmill technique, a manual removal is performed according to the clinic standard.
  Interventions: Other: Windmill at 30 Minutes
- Control Group (Active Comparator): In the control group, after a total of 45 minutes of unsuccessful application of the traditional and customary measures, the Windmill technique is used. If unsuccessful, a manual placenta removal is performed according to hospital Standards.
  Interventions: Other: Windmill at 45 Minutes

INTERVENTIONS:
Other: Windmill at 30 Minutes — The so-called windmill technique of placenta development for the management of the retained placenta involves the application of a continuous 360-degree umbilical traction force with centripetal rotation in such a way that it runs at the level of the introitus perpendicular to the direction of the birth canal. This rotation around a 360-degree traction plane is repeated slowly and continuously with a motion that resembles the motion of the wings of a windmill until the placenta can be safely delivered.
  Arms: Windmill group 30 Mins
Other: Windmill at 45 Minutes — The so-called windmill technique of placenta development for the management of the retained placenta involves the application of a continuous 360-degree umbilical traction force with centripetal rotation in such a way that it runs at the level of the introitus perpendicular to the direction of the birth canal. This rotation around a 360-degree traction plane is repeated slowly and continuously with a motion that resembles the motion of the wings of a windmill until the placenta can be safely delivered.
  Arms: Control Group

SUMMARY:
The incidence of leftover placenta after vaginal delivery is between 0.1% and 3.3%, with a maternal mortality of up to 10% reported. The traditional management is ultimately the manual removal of the retained placenta (MROP) in the operating room. However, MROP itself increases the risk of further bleeding, postpartum infection, uterine perforation and inversion of the uterus. In a preliminary study with a small cohort, the "Windmill Technique" has already been successfully tested.

DETAILED DESCRIPTION:
The Windmill technique of placenta development for the management of the retained placenta involves the application of a continuous 360-degree umbilical traction force with centripetal rotation in such a way that it runs at the level of the introitus perpendicular to the direction of the birth canal.

The aim of this prospective randomized study is to compare the Windmill placental development technique with traditional placental development strategies. It also analyzes the need to carry out MROP in both groups.

The primary objective of the study is to compare the success rate of removing the placenta in retained placenta pregnancies between the Windmill technique and the control group. Based on this objective, we expected the difference of success rate between groups of 30% (from the previous study, the success rate of the Windmill technique was 86%]. The sample size of 35 participants per group will be required to provide 90% power at a 0.05 two-sided significance level.

ELIGIBILITY:
Inclusion Criteria:

* Presence of the written consent of the patient
* The patients must be over 18 years old
* Patients are not limited in their ability to consent

Exclusion Criteria:

* Age under 18
* Limited ability to work
* Known coagulation disorder
* Blood loss> 500ml
* Known placenta accreta
* No extension of the umbilical cord on traction.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Delivery of the placenta | At the end of delivery
  Successful delivery of the placenta

SECONDARY OUTCOMES:
Need for Manual Removal of Placenta | At the end of delivery
  Operative manual removal of placenta
Blood loss | At the end of delivery
  Estimated and Calculated Blood Loss

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Hospital, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hinkson L, Suermann MA, Hinkson S, Henrich W. The Windmill technique avoids manual removal of the retained placenta-A new solution for an old problem. Eur J Obstet Gynecol Reprod Biol. 2017 Aug;215:6-11. doi: 10.1016/j.ejogrb.2017.05.028. Epub 2017 Jun 1. PMID 28591673